CLINICAL TRIAL: NCT01514604
Title: Constructing a Learning Curve in Ultrasound Guided Needling - an Observational Study Using Cumulative Sum (Cusum) Analysis
Brief Title: Constructing a Learning Curve in Ultrasound Guided Needling
Status: Completed | Type: Observational
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Other Study IDs: 11/NS/0040
Record Dates: First submitted 2012-01-17; First posted 2012-01-23 (Estimated); Last update posted 2014-04-30 (Estimated); Status verified 2014-04

CONDITIONS: In-plane Ultrasound Guided Needling Training
Keywords: Anesthesia and analgesia; ultrasonography; education
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Little or no experience.: All participants will be asked to declare their degree of experience in the technique being studied. Those declaring themselves as 'New to in-plane ultrasound guided needling. Little or no experience in technique' belong to this cohort and will form the study group.
- Regular practitioner. Teaching: Participants declaring themselves as 'Regularly incorporate in-plane ultrasound guided needling in clinical practice. Teaching technique to others' fall within this cohort and form the 'control' group allowing application of a realistic acceptable failure rate to Cusum analysis of the study group.
- Some exposure. Infrequent clinical use.: Participants declaring themselves as belonging to this group will not form part of the analysis. They will be welcome to complete training and receive feedback on their performance according to the study protocol.

SUMMARY:
Constructing a learning curve in ultrasound guided needling

Observational study - How many attempts, with continuous training and feedback, at in-plane ultrasound guided needling in a phantom model are required to attain competence?

The use of ultrasound to enable real-time needle visualisation during regional anaesthesia (placing local anaesthetic, via a needle, near nerves to result in numbing of an area of the body to be operated on) has gained in popularity in recent years. It has been recognised by NICE (National Institute for Clinical Excellence) and guidelines on training have been published, with UK equivalents pending. These call for training in the technique on models or 'phantoms' prior to patient contact.

It is unknown how much experience is necessary to attain competence in a phantom, prior to proceeding to patient contact. One study looking at experiential learning of the technique found a very wide range of experience needed between individuals.

In order to study the effect of any changes in training methods on the learning of the technique it is necessary to have a baseline learning curve.

The investigators are introducing a training package for anaesthetists new to the technique to meet the recommendations on initial phantom based training. Alongside this the investigators aim to gather prospective observational data allowing the investigators to generate a learning curve for the technique. This involves making a video recording of the ultrasound images of approximately 50 sequential attempts at performing a task in a phantom, with ongoing instruction and coaching. The whole training package will take approximately 1 hour.

These video clips will be reviewed and sequential attempts graded for quality of needle visualisation and task completion. This will allow the investigators to use a statistical method, Cumulative Sum (Cusum) analysis, to determine how many attempts were required to attain proficiency. The investigators hope to recruit approximately 20 participants to this pilot study, and from this determine the average amount of training necessary to attain proficiency. Using Cusum analysis requires the use of an acceptable failure rate, usually chosen arbitrarily. To add greater meaning to our findings the investigators will also invite anaesthetists experienced in the technique of in-plane ultrasound guided needling to participate. By measuring the actual success rate of our local trainers the investigators will be able to make a meaningful comparison of the training required to achieve a similar level of success.

DETAILED DESCRIPTION:
1.0 INTRODUCTION

1.1 BACKGROUND INFORMATION

The use of ultrasound as a tool for guiding regional anaesthesia has been growing in popularity and use. The National Institute of Clinical Excellence (NICE) has acknowledged the role of ultrasound in regional anaesthesia by issuing guidance governing incorporation in clinical practice. The focus of this guidance was on the adoption of ultrasound by properly trained practitioners in a setting of adequate clinical governance, consent and audit. [1] Trainees in anaesthesia are expected to become familiar with regional anaesthetic techniques, increasingly involving the use of ultrasound. Of paramount importance is the acquisition of the skill of needle visualisation under ultrasound guidance in real time. There is growing consensus that trainees should undergo a period of training on a phantom prior to performing techniques on patients [2, 3].

Given the increasing use of ultrasound for regional anaesthesia within our trust, together with the recognition of the requirement for adequate formal training in its use we plan to introduce a program of phantom based training in ultrasound needle visualisation and control for trainees prior to commencing clinical practice.

1.2 RATIONALE FOR CURRENT STUDY

The amount of training required to achieve competency, both on phantom models or in clinical practice is unknown. Some work has been done using the cumulative sum (CUSUM) method with several different anaesthetic related practical procedures. These show that individual learning curves vary greatly, however the CUSUM method has shown promise as a technique for determining the acquisition of competence. [4, 7] Unsurprisingly it has also been suggested that providing training, before and during phantom practice, improves the success and rate of skill acquisition [4, 5, 6]. In order to conduct any future work into the effect of interventions in training methods on learning curves in regional anaesthesia a baseline learning curve needs to be constructed. As part of our planned training program we intend to collect observational data to enable the construction of a baseline learning curve for the attainment of competence in ultrasound needle visualisation.

One of the weaknesses of previous attempts at incorporating CUSUM into training analysis has been the need to arbitrarily select values for acceptable and unacceptable failure rates. We hope to address this in our study by simultaneously determining the local failure rate of the technique amongst proficient practitioners, and applying this data in CUSUM analysis of data collected during novice training. In order to provide pragmatic data applicable to the average anaesthetic department we will define proficient practitioners, for the purposes of calculating acceptable failure rates, as those anaesthetists routinely incorporating in-plane ultrasound guided needle visualisation in their practice and teaching it to others.

The investigators suggest that providing novices with instruction during the practice process, rather than allowing a 'discovery learning' approach as previously studied [4], will result in a lower total and narrower spread of attempts required to attain competence. By using a measured acceptable failure rate we will add validity to our data.

2. STUDY OBJECTIVES

Primary objective - Determine the amount of training required (number of attempts) to attain statistical proficiency in the average anaesthetist.

Secondary outcomes - Determine the effect of prior experience or demographic factors on the rate of skill acquisition.

Determine whether trainer assessment predicts statistical outcome.

3. STUDY DESIGN

The proposed study will be a prospective observational study.

We aim to recruit 20 participants in this pilot study.

Methods -

Anaesthetists within the department will be invited to participate in a short training and observational exercise.

Participants will be asked for consent in advance to have the ultrasound images of their practice attempts recorded anonymously and subsequently assessed. Refusal of consent will not preclude them from taking part in the training if desired.

Participants will be asked to provide some background demographic data on subjects which may be expected to effect the rate of skill acquisition. This will include age, sex, grade of anaesthetist, prior experience with in-plane ultrasound guided needling (regional anaesthesia or vascular access), exposure to computer gaming. (See Appendix)

Participants will be asked to declare their level of experience

1. New to in-plane ultrasound guided needling. Little or no experience in technique.
2. Some exposure to in-plane ultrasound guided needling. Infrequent use in clinical practice.
3. Regularly incorporate in-plane ultrasound guided needling in clinical practice. Teaching technique to others.

   Experience gained in Ultrasound Guided Regional Anaesthesia and vascular access techniques will be deemed valid.

   All participants, irrespective of previous experience, will then complete a training / observational package as detailed below.

   Training sessions will be run on a one to one basis by the local Fellow in Regional Anaesthesia. Participants will spend approximately 15 minutes viewing a brief powerpoint presentation introducing the principles of ultrasound followed by machine orientation and instruction on needle handling and visualisation techniques. The trainer will demonstrate the technique.

   Participants will then spend approximately 45 minutes of hands on practice at needle handling and visualisation while performing a task in a standardised gelatin based phantom. Instruction and feedback will be provided throughout, with the aim being to develop or demonstrate skill in maintaining needle tip visualisation at all times while advancing towards and contacting a target. It is anticipated that participants will undertake approximately 50 needle passes during this time.

   For each attempt the participant will be asked to advance the needle under ultrasound guidance toward a target, maintaining constant needle visualisation to the best of their ability. A brief period of initial shallow insertion to locate the needle with ultrasound will be permitted, as will partial withdrawal and re-alignment of the needle. A fresh puncture of the phantom will be regarded as the next attempt. Once participants feel they have optimised the needle position contacting the target the trainer will ensure optimal needle visualisation to exclude tip placement within or traversing the target. The needle will be withdrawn and the participant proceeds to the next attempt.

   We will be using a Sonosite M-Turbo ultrasound machine with HFL38X 6-13MHz linear probe and Sonoplex 80mm 20G needles. Ultrasound images will be recorded digitally using an "iGrabber" USB video capture device onto a laptop computer. Recording will start immediately prior to needle insertion. Once the participant has optimised needle position for that attempt the image will be frozen to indicate the end point, unfrozen and visualisation of the needle optimised by the trainer (with participant maintaining static needle position) before withdrawal of the needle, after which recording will be stopped. The process will be repeated for each subsequent attempt. At the end of the period of training of participants rating themselves as within group 1 the trainer will record whether they feel the participant has demonstrated competence, for later comparison with CUSUM analysis.

   Following this period of training and observation the anonymised video recordings of the participants attempts will be exported for review by two consultant anaesthetists, each experienced in ultrasound guided regional anaesthesia. Each needle pass will be assessed, out of sequence, and graded against previously agreed criteria based on a previously published system [4](appendix). Sequential grading information for each participant will be collated. Data for participants in group 3 will be used to calculate the actual failure rate of anaesthetists within our department considering themselves competent enough to teach the technique. This will be used as the acceptable failure rate to generate a CUSUM chart for those participants in group 1 to assess the attainment of competence. If desired this information will subsequently be fed back to the participant, but will not play any part in determining the progress of their training or practice.

   3.1 STUDY OUTCOME MEASURES

   The outcome will be an indication of the amount of training required to attain competence in the average novice anaesthetist, validated by using the measured success rate of those already deemed competent working within the department.
4. PARTICIPANT ENTRY

   4.1 PRE-REGISTRATION EVALUATIONS Nil

   4.2 INCLUSION CRITERIA Any anaesthetist within the anaesthetic dept of Aberdeen Royal Infirmary or Woodend Hospital, Aberdeen providing written, informed consent.

   4.2 EXCLUSION CRITERIA Refusal of consent.

   4.3 WITHDRAWAL CRITERIA Participants are free to withdraw from the study at any time, with no detriment to training offered.
5. ASSESSMENT AND FOLLOW UP

   Following construction of CUSUM charts and analysis of each participants performance, the individuals results will be fed-back to them if desired. No further follow-up is planned beyond this. Following feedback links between data and person-identifiable information will be broken.
6. STATISTICS AND DATA ANALYSIS

   This is a pilot project and a power calculation was not possible.

   Assistance will be given by the medical statistics department of the University of Aberdeen with the construction of CUSUM charts and any subsequent analysis if required.
7. REGULATORY ISSUES

7.1 ETHICS APPROVAL

The Chief Investigator will obtain ethics approval from the North of Scotland Regional Ethics Committee. The study will be submitted for Site Specific Assessment (SSA) at each participating NHS Trust. The Chief Investigator will require a copy of the SSA approval letter before accepting participants into the study. The study will be conducted in accordance with the recommendations for physicians involved in research on human subjects adopted by the 18th World Medical Assembly, Helsinki 1964 and later revisions.

7.2 CONSENT

All potential participants will be provided invitation and participant information letters detailing the study aims, objectives and protocol. A minimum period of overnight will be allowed to peruse information, after which an opportunity to discuss the study will be made available prior to seeking informed, written consent. An independent point of contact will be available to discuss the study if desired. Participants are free to cease participation in the study at any point if desired, with no effect on training opportunity. Equally should potential participants refuse consent to the study, they may complete the training session if desired.

7.3 CONFIDENTIALITY

The Chief Investigator will preserve the confidentiality of the participants taking part in the study.

All data will be collected under an individual study number only. A separate database will be held linking participant contact details to study numbers. To further decrease the possibility of participant identification by assessors video clips will be assessed in batches of five.

Following feedback of statistical performance to participants links between data and person-identifiable information will be broken.

All data will be collected in paper form then transferred to a digital format. Paper copies will be stored in a locked box in the acute pain team office at woodend hospital. Digital information will be stored on a password protected account on the NHS Grampian computer network.

It will be necessary to process the anonymised video recordings on a home computer prior to assessment.

ELIGIBILITY:
Inclusion Criteria:

* Any anaesthetist working within the anaesthetic dept of Aberdeen Royal Infirmary or Woodend Hospital, Aberdeen providing written, informed consent.

Exclusion Criteria:

* Refusal of consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Anaesthetists working within the anaesthetic department of Aberdeen Royal Infirmary / Woodend hospitals, Aberdeen.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2012-03; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Attempts required to achieve proficiency as assessed by CUSUM analysis, using data from actual local failure rate. | 1 year

SECONDARY OUTCOMES:
Relationship between demographic factors or prior experience and the primary outcome | 1 year
  We will record data including gender, grade of anaesthetist, prior exposure to ultrasound guided needling and prior video gaming experience and relate this to attainment of statistical competency during the training and observation.
Relationship between trainers impression of competence and statistical competence? | 1 year
  Trainers will be asked to record their impression of whether a participant has demonstrated competency following training, prior to scoring and analysis of the video recordings. We will compare the trainers impression with the outcome of scoring and cusum analysis for each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Bourke, MBChB. FRCA, Principal Investigator — NHS Grampian
Locations (1):
- Aberdeen Royal Infirmary / Woodend Hospital, Aberdeen, Aberdeenshire, United Kingdom